CLINICAL TRIAL: NCT02912195
Title: Intravenous Lidocaine Versus Provider Chosen Dose of Morphine for the Treatment of Severe Pain in the Emergency Department: An Open-label Randomized Controlled Pilot Study
Brief Title: Intravenous Lidocaine Versus Morphine for Severe Pain in the ED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alameda Health System (Other)
Responsible Party: Principal Investigator, Eben Clattenburg, Principle Investigator, Alameda Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00001
Record Dates: First submitted 2016-09-20; First posted 2016-09-23 (Estimated); Results first posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous lidocaine (Experimental): Participants will receive IV lidocaine (75 mg if <50kg, 100 mg if 50 - 100 kg, and 150 mg if >100 kg) over 10 minutes in a 100 mL normal saline minibag followed by a 50 minute IV lidocaine drip (75 mg if <50kg, 100 mg if 50 - 100 kg, and 150 mg if >100 kg) in a 100 mL normal saline minibag.
  At 20 and 40 minutes, participants can elect to receive morphine 4mg IV as a rescue analgesic.
  Interventions: Drug: Intravenous lidocaine
- Morphine (Active Comparator): ED provider will choose an appropriate dose of intravenous morphine for the patient.
  At 20 and 40 minutes, participants can elect to receive morphine 4mg IV as a rescue analgesic.
  Interventions: Drug: Intravenous morphine

INTERVENTIONS:
Drug: Intravenous lidocaine — Intravenous lidocaine drip over 10 minutes followed by intravenous lidocaine drip over 50 minutes
  Other Names: lignocaine; Xylocaine
  Arms: Intravenous lidocaine
Drug: Intravenous morphine — Emergency department provider chooses appropriate dose of intravenous morphine
  Other Names: duramorph
  Arms: Morphine

SUMMARY:
Objective: Evaluate the analgesic efficacy of intravenous (IV) lidocaine versus provider chosen dose of IV morphine for the treatment of severe pain in the emergency department.

Study design: Open-label, randomized controlled pilot study.

DETAILED DESCRIPTION:
Objective: The purpose of this pilot study is to determine the analgesic efficacy of intravenous lidocaine versus morphine for the treatment of severe pain in the emergency department (ED).

Study design: Open-label, randomized, controlled pilot trial. Participants: Investigators and research assistants will recruit patients ≥18 years old with severe pain (NRS ≥7) and an anticipated stay in the emergency department ≥1 hour. A sample size calculation was performed and 32 patients will be enrolled.

Intervention: After a trained research assistant obtains written informed consent, eligible participants will be randomized to the intravenous lidocaine or morphine arms of the study. In the intravenous lidocaine arm, patients will receive IV lidocaine (75 mg if <50kg, 100 mg if 50 - 100 kg, and 150 mg if >100 kg) over 10 minutes in a 100 mL normal saline minibag followed by a 50 minute IV lidocaine drip (75 mg if <50kg, 100 mg if 50 - 100 kg, and 150 mg if >100 kg). In the morphine arm, the ED provider will choose an appropriate dose of morphine for the patient. At 20 and 40 minutes, the participants will be asked "Would you like additional pain medication?". Participants responding in the affirmative will receive morphine 4 mg IV.

Data collection: The trained research assistant will collect data on the patients' pain scores, side effects, and rescue morphine.

Statistical analysis: Investigators will perform descriptive statistics and compare pain scores and pain relief at each time point with unpaired t-tests.

ELIGIBILITY:
Inclusion Criteria:

* Subject has severe pain (NRS ≥7)
* Subject has anticipated ED stay of ≥1 hour

Exclusion Criteria:

* High acuity trauma patients
* Patients deemed to critically ill by ED provider
* Active psychosis
* Pregnancy
* History of heart block or bradycardia
* Allergy to lidocaine or amide type local anesthetic
* History of seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Herring, MD, Principal Investigator — Alameda Health System, Highland Hospital
Locations (1):
- Alameda Health System, Highland Hospital, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous Lidocaine: Participants will receive IV lidocaine (75 mg if <50kg, 100 mg if 50 - 100 kg, and 150 mg if >100 kg) over 10 minutes in a 100 mL normal saline minibag followed by a 50 minute IV lidocaine drip (75 mg if <50kg, 100 mg if 50 - 100 kg, and 150 mg if >100 kg) in a 100 mL normal saline minibag.
  At 20 and 40 minutes, participants can elect to receive morphine 4mg IV as a rescue analgesic.
  Intravenous lidocaine: Intravenous lidocaine drip over 10 minutes followed by intravenous lidocaine drip over 50 minutes
- Morphine: ED provider will choose an appropriate dose of intravenous morphine for the patient.
  At 20 and 40 minutes, participants can elect to receive morphine 4mg IV as a rescue analgesic.
  Intravenous morphine: Emergency department provider chooses appropriate dose of intravenous morphine
Period: Overall Study
Arm/Group | Intravenous Lidocaine | Morphine
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Lidocaine | Morphine | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [36.5 to 59.5] | 45.5 [34 to 59.5] | 46 [36 to 59.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 8 | 7 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pain Score (NRS 0-10)
Description: Pain score is rated on the Numeric Rating Scale from 0-10. 0 represents no pain and 10 represents the worst possible pain.
Time Frame: At 60 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intravenous Lidocaine | Morphine
Number analyzed (Participants) | 16 | 16
units on a scale | 5.1 [3.3 to 6.8] | 4.2 [3.0 to 5.4]

2. Secondary Outcome: Pain Score (NRS 0-10)
Description: Pain score recorded on the numeric rating scale 0-10.
Time Frame: At 10 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intravenous Lidocaine | Morphine
Number analyzed (Participants) | 16 | 16
units on a scale | 8.1 [7.1 to 9.0] | 8.9 [8.3 to 9.6]

3. Secondary Outcome: Pain Score (NRS 0-10)
Description: Pain score recorded on the numeric rating scale 0-10. 0 represents no pain and 10 represents the worst pain.
Time Frame: At 20 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intravenous Lidocaine | Morphine
Number analyzed (Participants) | 16 | 16
units on a scale | 7.4 [6.3 to 8.4] | 6.2 [4.6 to 7.8]

4. Secondary Outcome: Pain Score (NRS 0-10)
Description: Pain score recorded on the numeric rating scale 0-10.
Time Frame: At 30 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intravenous Lidocaine | Morphine
Number analyzed (Participants) | 16 | 16
units on a scale | 7.0 [5.9 to 8.1] | 5.6 [4.0 to 7.1]

5. Secondary Outcome: Pain Score (NRS 0-10)
Description: Pain score recorded on the numeric rating scale 0-10.
Time Frame: At 40 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intravenous Lidocaine | Morphine
Number analyzed (Participants) | 16 | 16
units on a scale | 6.3 [5.0 to 7.5] | 4.7 [3.2 to 6.3]

6. Secondary Outcome: Pain Score (NRS 0-10)
Description: Pain score recorded on the numeric rating scale 0-10.
Time Frame: At 50 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intravenous Lidocaine | Morphine
Number analyzed (Participants) | 16 | 16
units on a scale | 5.6 [4.1 to 7.1] | 4.6 [3.1 to 6.0]

7. Secondary Outcome: Pain Relief at 10 Minutes Compared to Baseline.
Description: Pain NRS at 0 minutes minus pain NRS at 10 minutes
Time Frame: At 10 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intravenous Lidocaine | Morphine
Number analyzed (Participants) | 16 | 16
units on a scale | 1.1 [0.5 to 1.8] | 2.0 [0.9 to 3.0]

8. Secondary Outcome: Pain Relief at 20 Minutes Compared to Baseline.
Description: Pain numeric rating scale (NRS) at 0 minutes minus pain NRS at 20 minutes. NRS is a scale ranging from 0, no pain, to 10 worst pain.
Time Frame: at 20 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intravenous Lidocaine | Morphine
Number analyzed (Participants) | 16 | 16
units on a scale | 1.8 [1.1 to 2.5] | 2.8 [1.4 to 4.1]

9. Secondary Outcome: Pain Relief at 30 Minutes Compared to Baseline.
Description: Pain numeric rating scale (NRS) at 0 minutes minus pain NRS at 30 minutes NRS is a scale ranging from 0, no pain, to 10 worst pain.
Time Frame: at 30 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intravenous Lidocaine | Morphine
Number analyzed (Participants) | 16 | 16
units on a scale | 2.2 [1.4 to 3.0] | 3.4 [1.9 to 4.7]

10. Secondary Outcome: Pain Relief at 40 Minutes Compared to Baseline.
Description: Pain numeric rating scale (NRS) at 0 minutes minus pain NRS at 40 minutes. NRS is a scale ranging from 0, no pain, to 10 worst pain.
Time Frame: At 40 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intravenous Lidocaine | Morphine
Number analyzed (Participants) | 16 | 16
units on a scale | 2.9 [1.7 to 4.1] | 4.2 [2.9 to 5.6]

11. Secondary Outcome: Pain Relief at 50 Minutes Compared to Baseline.
Description: Pain numeric rating scale (NRS) at 0 minutes minus pain NRS at 50 minutes. NRS is a scale ranging from 0, no pain, to 10 worst pain.
Time Frame: At 50 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intravenous Lidocaine | Morphine
Number analyzed (Participants) | 16 | 16
units on a scale | 3.6 [2.2 to 5.0] | 4.4 [3.2 to 5.6]

12. Secondary Outcome: Pain Relief at 60 Minutes Compared to Baseline.
Description: Pain numeric rating scale (NRS) at 0 minutes minus pain NRS at 60 minutes. NRS is a scale ranging from 0, no pain, to 10 worst pain.
Time Frame: At 60 minutes
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Intravenous Lidocaine | Morphine
Number analyzed (Participants) | 16 | 16
units on a scale | 4.1 [2.6 to 5.7] | 4.8 [3.7 to 5.8]

13. Secondary Outcome: Number of Participants Requiring Rescue Medications
Description: The percentage of patients requiring rescue IV morphine at 20 and 40 minutes
Time Frame: At 20 and 40 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Lidocaine | Morphine
Number analyzed (Participants) | 16 | 16
Participants | 5 | 4

14. Secondary Outcome: Patient Satisfaction
Description: The proportion of patients saying, "Yes" to "Would you have this pain medication again for similar pain?"
Time Frame: 60 minutes
Population: 1 patient in the intravenous lidocaine arm did not answer the question.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Lidocaine | Morphine
Number analyzed (Participants) | 15 | 16
Participants | 13 | 14

15. Secondary Outcome: Number of Participants Reporting Adverse Events
Description: Participants will be observed for the following adverse events and side effects: seizure, bradyarrhythmias, hyper or hypotension, perioral numbness, tinnitus, metallic taste, other, hypotension, hypoxia, nausea, vomiting, itching, or other side effects. Participants have the opportunity to report other side effects during the study
Time Frame: 0-60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Lidocaine | Morphine
Number analyzed (Participants) | 16 | 16
Participants | 2 | 6

ADVERSE EVENTS:
Arm/Group | Intravenous Lidocaine | Morphine
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/16 | 6/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Lidocaine (N=16) | Morphine (N=16)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Perioral numbness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
bradycardia (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was limited by a small sample size and lack of blinding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No